CLINICAL TRIAL: NCT04450342
Title: A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Efficacy of ARCR Augmented With REGENETEN™ Bioinductive Implant System in Full-thickness Tears (Large or Massive) Repair Versus ARCR Alone
Brief Title: REGENETEN™ Bioinductive Implant System in Full-thickness Tears
Acronym: REGENETEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision not related to safety.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REGENETEN.2020.01
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2023-11

CONDITIONS: Rotator Cuff Injuries
Keywords: Rotator cuff tendon; Full thickness tears; REGENETEN Bioinductive Implant System
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Reoperation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- ARCR augmented with REGENETEN™ Bioinductive Implant (Experimental): During the ARCR procedure, the REGENETEN™ Bioinductive Implant is covering the tendon and attached to the bone and the tendon with small anchors.
  Interventions: Device: Arthroscopic rotator cuff repair with REGENETEN™ Bioinductive Implant augmentation
- ARCR alone (Sham Comparator): The rotator cuff is repaired during arthroscopic standard procedure. No product is added for healing
  Interventions: Procedure: Arthroscopic rotator cuff repair
- Revision group (Other): Revision group allows treatment of subjects having recurrent tears, ARCR supplemented with REGENETEN
  Interventions: Device: Arthroscopic rotator cuff repair for revision surgery

INTERVENTIONS:
Device: Arthroscopic rotator cuff repair with REGENETEN™ Bioinductive Implant augmentation — The Arthroscopic rotator cuff repair aims at repairing the rotator cuff following tendon tear. The REGENETEN Bioinductive Implant is a medical device intended for the management and protection of tendon injuries. The REGENETEN Bioinductive Implant is indicated for the management and protection of rotator cuff tendon injuries in which there has been no substantial loss of tendon tissue. The REGENETEN Bioinductive Implant is a bioabsorbable implant device that provides a layer of collagen over injured tendons. The implant is designed to provide a layer of collagen between a flat tendon and the surrounding tissue. After hydration, the implant is an easy-to-handle, pliable, nonfriable, porous collagen sheet.
  Arms: ARCR augmented with REGENETEN™ Bioinductive Implant
Procedure: Arthroscopic rotator cuff repair — The Arthroscopic rotator cuff repair aims at repairing the rotator cuff following tendon tear without supplement.
  Arms: ARCR alone
Device: Arthroscopic rotator cuff repair for revision surgery — The Arthroscopic rotator cuff repair can also occur in recurrent tears. The REGENETEN Bioinductive Implant will be applied during the ARCR procedure.
  Arms: Revision group

SUMMARY:
The study is designed to assess the safety and efficacy of Arthroscopic rotator cuff repair (ARCR) augmented with REGENETEN in subjects requiring full-thickness rotator cuff tear repair or revision repair versus Arthroscopic rotator cuff repair alone.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized, controlled clinical study in the treatment of full thickness tears of the rotator cuff (large or massive ≥3 cm in AP or ML according to Cofield classification). The subjects meeting the inclusion/exclusion criteria specified in the protocol will receive either ARCR augmented with REGENETEN or ARCR alone. Subjects enrolled into the revision repair subject group will receive ARCR augmented with REGENETEN. The clinical follow-up evaluation will be performed preoperatively (Baseline), 2 weeks, 6 weeks, 3, 6, 12, and 24 months after surgery, respectively using subjective outcome measures, objective measures of movement and an MRI scan to assess the integrity of the repair and assess the re-tear rate. Health economic data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Subject requires Arthroscopic rotator cuff repair (ARCR);
2. Subjects with a diagnosis of a symptomatic primary or recurrent (revision repair subject group), large or massive tear (≥ 3 cm AP/ML) of the supraspinatus and/or infraspinatus tendons amenable to repair. For screening purposes, a ≥ 2 cm AP/ML tear as measured on MRI will be eligible to proceed to the operative visit but will have to be confirmed as ≥ 3 cm on arthroscopy using a calibrated probe to proceed;
3. Subject is > 40 years of age (no upper limit);
4. Subject provides written informed consent for study participation using an Independent Ethical Committee (IEC) / Institutional Review Board (IRB) approved consent form;
5. Subject is willing and able to participate in required follow-up visits and is able to complete study activities.

Exclusion Criteria:

1. Subjects who are unable to tolerate magnetic resonance imaging (MRI), due to psychiatric or medical contraindications;
2. Subjects with Samilson-Prieto osteoarthritis > 2;
3. Subjects with current or prior infection of the ipsilateral shoulder;
4. Subjects with known hypersensitivity to bovine-derived materials;
5. Subjects with known inflammatory arthropathy, history of inflammatory arthropathy, or chronic joint disease;
6. Subjects with prior shoulder surgery (not including rotator cuff repair [revision repair subject group only], biceps tenodesis/tenotomy, distal clavicle excision [DCE], subacromial decompression);
7. Subjects with an irreparable or partially reparable rotator cuff tear;
8. Subjects with a subscapularis tear requiring repair;
9. Subjects requiring a concomitant labral fixation procedure;
10. Subjects requiring a concomitant os acromiale fixation procedure;
11. Subjects with glenohumeral joint instability (multiple dislocations/subluxations);
12. Subjects with a subacromial or intra-articular injection within 3 months prior to surgery;
13. Subjects with condition(s) that contraindicate or complicate outcomes of ARCR e.g., > Hamada 3 rotator cuff arthropathy on X-ray, Goutallier atrophy > Grade 3, proximal humeral fracture or scapular fracture, avascular necrosis of the humeral head or glenoid, history of immunodeficiency disorders, history of chronic inflammatory disorders, oral or injected steroid use in last 4 weeks;
14. Subjects who are pregnant or breast feeding;
15. Subjects who are currently involved in any injury litigation or workers compensation claims;
16. Subjects who are enrolled, or plan to enroll, in another clinical trial during this study that would affect the outcomes of this study;
17. Subjects with a history of noncompliance with medical treatment, physical therapy (PT)/rehabilitation, or clinical study participation
18. Subject who, in the opinion of the Investigator, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, and drug or alcohol abuse;
19. Subjects who do not meet the indication or are contraindicated according to specific Smith+Nephew REGENETEN System's Instructions for Use (IFUs);
20. Subject that meets the definition of a Vulnerable Subject per ISO14155:2020 Section 3.44.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Peach, MBBS MD FRCS (Tr&Orth), Principal Investigator — Manchester University NHS Foundation Trust
Locations (30):
- United States (8):
  - Harbin Clinic, Rome, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Sinai Hospital, Baltimore, Maryland
  - Syracuse Orthopedic Specialists, DeWitt, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Orthopedic Specialists, Bedford, Texas
  - Houston Methodist The Woodlands, The Woodlands, Texas
  - Ashland Memorial Medical Center, Ashland, Wisconsin
- Australia (2):
  - Macquarie University Hospital, Sydney, New South Wales
  - OrthoSport Victoria, Richmond, Victoria
- Canada (3):
  - Saint John Orthopaedics, Saint John, New Brunswick
  - McMaster University, Hamilton, Ontario
  - Women's College Hospital Toronto, Toronto, Ontario
- France (5):
  - Hôpital Ambroise Paré, Paris, Boulogne-Billancourt
  - Hôpital Pasteur 2, Nice, Provence-Alpes-Côte d'Azur Region
  - Clinique Saint-Jean - Montpellier, Montpellier
  - Bichat Hospital, Paris
  - Hôpital Privé de l'Ouest Parisien, Trappes, Île-de-France Region
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Singapore General Hospital, Singapore, Singapore
- Switzerland (2):
  - Balgrist University Hospital, Zurich
  - Schulthess Klinik, Zurich
- United Kingdom (8):
  - Royal Blackburn Hospital, Blackburn, Lancashire
  - University Hospital of South Manchester NHS Foundation Trust, Wythenshawe, Manchester
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool, Merseyside
  - Royal National Orthopaedic Hospital NHS Trust, Stanmore, Middlesex
  - Nottingham University Hospital, Nottingham, Nottinghamshire
  - University Hospitals Coventry and Warwickshire, Coventry, Warwickshire
  - The Royal Orthopaedic Hospital NHS Foundation Trust, Birmingham, West Midlands
  - Southmead Hospital, Bristol

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 119 participants were enrolled to the study at 15 sites.
Period: Overall Study
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Started | 47 | 48 | 24
Completed | 10 | 14 | 12
Not Completed | 37 | 34 | 12
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Device not used | 1 | 0 | 0
Not completed — Withdrawal by Subject & Study Terminated by Sponsor | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Protocol Deviation | 0 | 1 | 0
Not completed — Reoperation | 1 | 1 | 0
Not completed — Screen Failures | 0 | 0 | 2
Not completed — Site Terminated by Sponsor | 1 | 1 | 1
Not completed — Study Terminated by Sponsor | 31 | 29 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) included all participants that received the study device with data collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group | Total
Number analyzed (Participants) | 47 | 48 | 24 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (7.6) | 62.2 (8.7) | 58.3 (9.2) | 61.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 5 | 42
  Male | 31 | 27 | 19 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 0 | 6
  Not Hispanic or Latino | 40 | 41 | 21 | 102
  Unknown or Not Reported | 3 | 5 | 3 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White / Caucasian | 43 | 37 | 22 | 102
  Race: Black / African American | 0 | 2 | 1 | 3
  Race: Asian Indian | 1 | 1 | 0 | 2
  Race: Chinese | 3 | 5 | 0 | 8
  Race: Japanese | 0 | 0 | 0 | 0
  Race: Korean | 0 | 0 | 0 | 0
  Race: Vietnamese | 0 | 0 | 0 | 0
  Race: Other Asian | 0 | 1 | 0 | 1
  Race: Aboriginal and Torres Strait Islander | 0 | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Other | 0 | 2 | 1 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Number of participants analyzed indicated those in the safety analysis set (SAF) with data collected for measure specified.
  kg/m^2
    number analyzed (Participants) | 45 | 46 | 24 | 115
    (all) | 29.7 (6.0) | 29.5 (5.8) | 28.3 (5.4) | 29.3 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Retear Rate at 6 Months
Description: Retear rate was measured by the percentage of retears 6 months after full-thickness arthroscopic rotator cuff repair (ARCR) surgery. Retear was defined as Sugaya Type IV or V retear/recurrence (full-thickness discontinuity seen on both coronal and oblique sagittal MRI images).
Time Frame: 6 months
Population: The full analysis set (FAS) followed the Intent-to-Treat principle that included participants enrolled into the study that attended at least one post-surgery assessment with data collected for the time frame and outcome indicated.
Measure: Number (95% Confidence Interval); unit: percentage of retears
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 42 | 19
percentage of retears | 57.14 [40.96 to 72.28] | 50.00 [34.19 to 65.81] | 42.11 [20.25 to 66.50]

2. Secondary Outcome: Number of Retears at 3 Months, 12 Months, and 24 Months
Description: Number of participants with retears present 3 months, 12 months, and 24 months after full-thickness arthroscopic rotator cuff repair (ARCR) surgery. Retear was defined as Sugaya Type IV or V retear/recurrence (full-thickness discontinuity seen on both coronal and oblique sagittal MRI images).
Time Frame: 3 months, 12 months, and 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 31 | 25 | 10
Participants
  3 months | 12 | 10 | 6
  12 months: number analyzed (Participants) | 13 | 9 | 0
  12 months | 7 | 6 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months | 1 | 1 |

3. Secondary Outcome: Oxford Shoulder Score (OSS)
Description: The Oxford Shoulder Score (OSS) is a questionnaire for the assessment of outcomes of shoulder surgery, which can reduce the observer's errors in the evaluation. It contains 12- item patient-reported outcome (PRO) measures specifically designed and developed for assessing outcomes of shoulder surgery such as assessing the impact on patients' quality of life of degenerative conditions (e.g., arthritis and rotator cuff problems). The OSS consists of 12 questions each scored 0 to 4 (0=unbearable, 1=severe, 2=moderate, 3=mild, 4=none) with 4 representing the best outcome. When the 12 items are summed, this produces overall scores that run from 0 to 48, with zero (0) representing a severe shoulder problem and 48 representing no related problem. Higher scores represent better clinical outcomes.
Time Frame: Baseline, 3 months, 6 months, 12 months and 24 months
Population: The full analysis set (FAS) followed the Intent-to-Treat principle that included participants enrolled into the study that attended at least one post-surgery assessment with data collected for the time frame and outcome indicated. Seven participants had out of range scores (i.e., scores were greater than the highest score possible) and were not included for analysis. No (0) Revision subjects completed the 12 or 24 month visit due to the early termination of the study or withdrawal of subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 44 | 45 | 23
score on a scale
  Baseline | 33.1 (7.7) | 34.0 (7.5) | 29.5 (7.8)
  3 months: number analyzed (Participants) | 32 | 29 | 14
  3 months | 25.1 (8.0) | 29.4 (9.7) | 23.4 (9.6)
  6 months: number analyzed (Participants) | 42 | 43 | 20
  6 months | 18.9 (6.6) | 19.9 (7.9) | 18.9 (7.6)
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months | 18.8 (8.5) | 17.3 (7.9) |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months | 19.0 (7.1) | 15.0 (4.2) |

4. Secondary Outcome: Western Ontario Rotator Cuff (WORC) / Chinese Version WORC (C-WORC) Index
Description: The WORC/C-WORC Index is self-administered, and includes a 5 different domains (physical symptoms, sports and recreation, work, social function, and emotions). Scores range from 0 to 2100 with 0 indicating no symptoms at all and 2100 indicating the worst possible symptoms (i.e., a lower score is a better outcome).
Time Frame: Baseline, 3 months, 6 months, 12 months and 24 months
Population: The full analysis set (FAS) followed the Intent-to-Treat principle that included participants enrolled into the study that attended at least one post-surgery assessment with data collected for the time frame and outcome indicated. No (0) Revision subjects completed the 12 or 24 month visit due to the early termination of the study or withdrawal of subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 46 | 48 | 24
score on a scale
  Baseline | 1271.3 (366.6) | 1307.5 (398.7) | 1194.0 (427.6)
  3 months: number analyzed (Participants) | 34 | 29 | 14
  3 months | 860.7 (350.1) | 936.7 (472.4) | 703.9 (365.1)
  6 months: number analyzed (Participants) | 43 | 43 | 20
  6 months | 533.6 (429.5) | 540.1 (475.1) | 548.8 (493.4)
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months | 432.8 (453.7) | 405.6 (596.5) |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months | 281.5 (252.4) | 62.5 (81.3) |

5. Secondary Outcome: Constant-Murley Score
Description: The Constant-Murley Score is a validated assessment of pain and shoulder functionality. The Constant Score is divided into 4 subscales: pain, activities of daily living, strength, and range of motion - forward flexion, external rotation, abduction and internal rotation of the shoulder. Scores range from 0 to 100 with a higher score indicating better shoulder function (i.e., a high score is a better outcome).
Time Frame: Baseline, 3 months, 6 months, 12 months and 24 months
Population: The full analysis set (FAS) followed the Intent-to-Treat principle that included participants enrolled into the study that attended at least one post-surgery assessment with data collected for the time frame and outcome indicated. Six participants had out of range scores (i.e., scores were greater than the highest score possible) and were not included for analysis. No (0) Revision subjects completed the 12 or 24 month visit due to the early termination of the study or withdrawal of subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 45 | 45 | 23
score on a scale
  Baseline | 56.5 (13.5) | 54.9 (13.7) | 55.6 (16.8)
  3 months: number analyzed (Participants) | 0 | 1 | 1
  3 months |  | 55.0 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 43.4 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis
  6 months: number analyzed (Participants) | 43 | 43 | 20
  6 months | 57.0 (13.0) | 53.7 (12.3) | 53.4 (9.4)
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months | 59.1 (13.8) | 57.2 (10.7) |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months | 58.5 (3.5) | 51.0 (11.3) |

6. Secondary Outcome: Subjective Shoulder Value (SSV)
Description: The Subjective Shoulder Value (SSV) is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder. The SSV ranges from 0 to 100, with a higher score indicating a better outcome.
Time Frame: Baseline, 3 months, 6 months, 12 months and 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 46 | 48 | 24
score on a scale
  Baseline | 38.3 (21.6) | 38.1 (24.6) | 47.1 (22.7)
  3 months: number analyzed (Participants) | 34 | 29 | 14
  3 months | 60.1 (21.0) | 57.1 (20.8) | 72.5 (16.8)
  6 months: number analyzed (Participants) | 43 | 43 | 20
  6 months | 74.1 (17.7) | 77.3 (20.6) | 76.3 (21.4)
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months | 80.0 (14.9) | 88.9 (10.2) |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months | 77.5 (24.7) | 91.5 (9.2) |

7. Secondary Outcome: EuroQol 5 Dimension 5 Level (EQ-5D-5L) Index Score
Description: The EQ-5D-5L score consists of two parts: a descriptive system and a visual analogue scale. The descriptive system is used to describe the participant's health state and consists of five dimensions to create an index score for mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas. The index score ranges from 0 to 1, with a higher score indicating a better outcome.
Time Frame: Baseline, 3 months, 6 months, 12 months and 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 46 | 48 | 24
score on a scale
  Baseline | 0.618 (0.186) | 0.574 (0.229) | 0.597 (0.216)
  3 months: number analyzed (Participants) | 34 | 29 | 14
  3 months | 0.720 (0.194) | 0.649 (0.206) | 0.776 (0.173)
  6 months: number analyzed (Participants) | 43 | 43 | 20
  6 months | 0.781 (0.216) | 0.786 (0.232) | 0.834 (0.165)
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months | 0.719 (0.227) | 0.805 (0.256) |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months | 0.679 (0.200) | 0.919 (0.115) |

8. Secondary Outcome: EuroQol 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale (VAS) Score
Description: The EQ-5D-5L score consists of two parts: a descriptive system and a visual analogue scale (VAS). The VAS score is the participant's self-rated health on a vertical visual analogue scale that ranges from 0 to 100 with 100 representing the best health imaginable and 0 indicating the worst (i.e., a higher score is a better outcome).
Time Frame: Baseline, 3 months, 6 months, 12 months and 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 46 | 48 | 24
score on a scale
  Baseline | 73.4 (15.4) | 69.8 (17.5) | 65.3 (23.1)
  3 months: number analyzed (Participants) | 34 | 29 | 14
  3 months | 74.2 (15.7) | 73.0 (16.4) | 80.3 (20.5)
  6 months: number analyzed (Participants) | 43 | 43 | 20
  6 months | 82.5 (15.4) | 79.3 (19.0) | 73.5 (21.8)
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months | 75.1 (16.6) | 75.0 (15.2) |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months | 30.0 (28.3) | 87.5 (3.5) |

9. Secondary Outcome: Patient Satisfaction Questionnaire: Medical Care
Description: The Patient Satisfaction Questionnaire was a simple subjective assessment from the patient's perspective for the question "How satisfied are you with your medical care?". Scores ranged from 0 to 100 with 0 indicating the least satisfied and 100 indicating the most satisfied.
Time Frame: Baseline, 3 months, 6 months, 12 months and 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 46 | 48 | 24
score on a scale
  Baseline | 88.6 (19.8) | 94.3 (8.3) | 89 (19.2)
  3 months: number analyzed (Participants) | 32 | 27 | 13
  3 months | 88.8 (13.7) | 93.1 (13.3) | 89.2 (27.3)
  6 months: number analyzed (Participants) | 39 | 41 | 19
  6 months | 89.7 (19.9) | 93.6 (16.6) | 90.8 (23.4)
  12 months: number analyzed (Participants) | 11 | 8 | 0
  12 months | 91.5 (11.3) | 94.4 (9) |
  24 months: number analyzed (Participants) | 1 | 1 | 0
  24 months | 90 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 90 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis |

10. Secondary Outcome: Patient Satisfaction Questionnaire: How Well Did the Surgery Relieve the Pain
Description: The post-operative Patient Satisfaction Questionnaire for pain relief was a simple subjective assessment from the patient's perspective at 3, 6, 12, and 24 months. Participants were asked to answer, "How well did the surgery relieve the pain?" with one of the following responses:
  * Excellent
  * Very Good
  * Good
  * Fair
  * Poor
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 43 | 20
Participants
  3 months: number analyzed (Participants) | 34 | 29 | 14
  3 months: Excellent | 7 | 9 | 5
  3 months: Very Good | 11 | 7 | 5
  3 months: Good | 11 | 4 | 1
  3 months: Fair | 3 | 6 | 2
  3 months: Poor | 2 | 3 | 1
  6 months: Excellent | 15 | 18 | 10
  6 months: Very Good | 17 | 13 | 6
  6 months: Good | 8 | 4 | 2
  6 months: Fair | 1 | 4 | 1
  6 months: Poor | 1 | 4 | 1
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months: Excellent | 5 | 6 |
  12 months: Very Good | 4 | 1 |
  12 months: Good | 1 | 1 |
  12 months: Fair | 0 | 1 |
  12 months: Poor | 2 | 0 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Excellent | 1 | 1 |
  24 months: Very Good | 0 | 1 |
  24 months: Good | 1 | 0 |
  24 months: Fair | 0 | 0 |
  24 months: Poor | 0 | 0 |

11. Secondary Outcome: Patient Satisfaction Questionnaire: How Well Did the Surgery Improve Your Ability to Perform Regular Activities
Description: The post-operative Patient Satisfaction Questionnaire for ability to perform regular activities was a simple subjective assessment from the patient's perspective at 3, 6, 12, and 24 months. Participants were asked to answer, "How well did the surgery improve your ability to perform regular activities?" with one of the following responses:
  * Excellent
  * Very Good
  * Good
  * Fair
  * Poor
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 43 | 20
Participants
  3 months: number analyzed (Participants) | 34 | 29 | 14
  3 months: Excellent | 5 | 1 | 1
  3 months: Very Good | 6 | 7 | 8
  3 months: Good | 14 | 6 | 1
  3 months: Fair | 4 | 9 | 2
  3 months: Poor | 5 | 6 | 2
  6 months: Excellent | 13 | 8 | 8
  6 months: Very Good | 16 | 21 | 6
  6 months: Good | 9 | 7 | 3
  6 months: Fair | 3 | 3 | 1
  6 months: Poor | 1 | 4 | 2
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months: Excellent | 5 | 6 |
  12 months: Very Good | 3 | 1 |
  12 months: Good | 2 | 2 |
  12 months: Fair | 1 | 0 |
  12 months: Poor | 1 | 0 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Excellent | 1 | 2 |
  24 months: Very Good | 0 | 0 |
  24 months: Good | 1 | 0 |
  24 months: Fair | 0 | 0 |
  24 months: Poor | 0 | 0 |

12. Secondary Outcome: Patient Satisfaction Questionnaire: How Well Did the Surgery Allow You to Perform Heavy Work or Sport Activities
Description: The post-operative Patient Satisfaction Questionnaire for performing heavy work or sport activities was a simple subjective assessment from the patient's perspective at 3, 6, 12, and 24 months. Participants were asked to answer, "How well did the surgery allow you to perform heavy work or sport activities?" with one of the following responses:
  * Excellent
  * Very Good
  * Good
  * Fair
  * Poor
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 41 | 43 | 20
Participants
  3 months: number analyzed (Participants) | 32 | 28 | 14
  3 months: Excellent | 0 | 1 | 1
  3 months: Very Good | 3 | 4 | 5
  3 months: Good | 10 | 1 | 2
  3 months: Fair | 9 | 9 | 3
  3 months: Poor | 10 | 13 | 3
  6 months: Excellent | 7 | 1 | 3
  6 months: Very Good | 10 | 20 | 6
  6 months: Good | 14 | 6 | 4
  6 months: Fair | 7 | 9 | 2
  6 months: Poor | 3 | 7 | 5
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months: Excellent | 2 | 5 |
  12 months: Very Good | 6 | 2 |
  12 months: Good | 1 | 1 |
  12 months: Fair | 2 | 1 |
  12 months: Poor | 1 | 0 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Excellent | 0 | 1 |
  24 months: Very Good | 1 | 1 |
  24 months: Good | 1 | 0 |
  24 months: Fair | 0 | 0 |
  24 months: Poor | 0 | 0 |

13. Secondary Outcome: Patient Satisfaction Questionnaire: How Well Did the Surgery Meet Your Expectations
Description: The post-operative Patient Satisfaction Questionnaire for surgery expectations was a simple subjective assessment from the patient's perspective at 3, 6, 12, and 24 months. Participants were asked to answer, "How well did the surgery meet your expectations?" with one of the following responses:
  * Excellent
  * Very Good
  * Good
  * Fair
  * Poor
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 43 | 20
Participants
  3 months: number analyzed (Participants) | 33 | 29 | 14
  3 months: Excellent | 11 | 8 | 8
  3 months: Very Good | 8 | 9 | 3
  3 months: Good | 9 | 7 | 0
  3 months: Fair | 4 | 3 | 1
  3 months: Poor | 1 | 2 | 2
  6 months: Excellent | 17 | 17 | 7
  6 months: Very Good | 11 | 13 | 5
  6 months: Good | 10 | 6 | 3
  6 months: Fair | 2 | 4 | 1
  6 months: Poor | 2 | 3 | 4
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months: Excellent | 5 | 6 |
  12 months: Very Good | 3 | 1 |
  12 months: Good | 1 | 2 |
  12 months: Fair | 2 | 0 |
  12 months: Poor | 1 | 0 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Excellent | 1 | 1 |
  24 months: Very Good | 0 | 1 |
  24 months: Good | 1 | 0 |
  24 months: Fair | 0 | 0 |
  24 months: Poor | 0 | 0 |

14. Secondary Outcome: Patient Satisfaction Questionnaire: Would You Have the Operation Again if Needed on Another Joint
Description: The post-operative Patient Satisfaction Questionnaire for having the operation again on another joint was a simple subjective assessment from the patient's perspective at 3, 6, 12, and 24 months. Participants were asked to answer, "Would you repeat the operation again if needed on another joint?" with one of the following responses:
  * Definitely Yes
  * Probably Yes
  * Possibly Not
  * Definitely Not
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 43 | 20
Participants
  3 months: number analyzed (Participants) | 34 | 29 | 14
  3 months: Definitely Yes | 20 | 18 | 11
  3 months: Probably Yes | 11 | 7 | 2
  3 months: Possibly Not | 2 | 0 | 1
  3 months: Definitely Not | 1 | 4 | 0
  6 months: Definitely Yes | 22 | 25 | 10
  6 months: Probably Yes | 14 | 12 | 7
  6 months: Possibly Not | 5 | 4 | 2
  6 months: Definitely Not | 1 | 2 | 1
  12 months: number analyzed (Participants) | 12 | 9 | 0
  12 months: Definitely Yes | 6 | 6 |
  12 months: Probably Yes | 3 | 1 |
  12 months: Possibly Not | 2 | 1 |
  12 months: Definitely Not | 1 | 1 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Definitely Yes | 2 | 1 |
  24 months: Probably Yes | 0 | 1 |
  24 months: Possibly Not | 0 | 0 |
  24 months: Definitely Not | 0 | 0 |

15. Secondary Outcome: Pain - Visual Analog Scale (VAS) Score
Description: Pain was measured using a 100-point Visual Analog Scale (VAS) score with a range from 0 to 100 where zero (0) represented no pain and 100 represented the worst pain imaginable (i.e., a lower score was a better outcome).
Time Frame: 2 weeks, 6 weeks, 3 months and 6 months
Population: The full analysis set (FAS) followed the Intent-to-Treat principle that included participants enrolled into the study that attended at least one post-surgery assessment with data collected for the time frame and outcome indicated. Data not collected for ARCR+Regeneten subjects at 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 43 | 42 | 24
score on a scale
  2 weeks | 31.2 (27.7) | 27.4 (26.6) | 21.6 (25.8)
  6 weeks: number analyzed (Participants) | 39 | 39 | 20
  6 weeks | 21.5 (24.3) | 24 (26.5) | 19.3 (23.8)
  3 months: number analyzed (Participants) | 0 | 1 | 1
  3 months |  | 20 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 2 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis
  6 months: number analyzed (Participants) | 21 | 24 | 13
  6 months | 10.4 (18) | 8 (17.9) | 9.2 (18.6)

16. Secondary Outcome: MRI Tendon Findings: Supraspinatus Sugaya Score
Description: The Sugaya Score was used to determine postoperative cuff integrity of the supraspinatus tendon through magnetic resonance imaging (MRI). Participants were classified as Type I, Type II, Type III, Type IV, Type V, or Indeterminate. Type I indicated sufficient thickness with homogenously low intensity. Type II indicates sufficient thickness with partial high intensity. Type III indicates insufficient thickness without discontinuity. Type IV indicates presence of a minor discontinuity, suggesting a small full-thickness tear. Type V indicates the presence of a major discontinuity, suggesting a medium or large full-thickness tear.
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: The safety analysis set (SAF) included participants that received the study device with data collected for the time frame and outcome indicated. Baseline score not collected as all participants had full-thickness tears. No (0) Revision subjects completed the 12 or 24 month visit due to the early termination of the study or withdrawal of subject.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 40 | 18
Participants
  3 months: number analyzed (Participants) | 31 | 25 | 9
  3 months: Type I | 1 | 0 | 0
  3 months: Type II | 17 | 15 | 3
  3 months: Type III | 1 | 0 | 0
  3 months: Type IV | 0 | 0 | 0
  3 months: Type V | 12 | 10 | 6
  3 months: Indeterminate | 0 | 0 | 0
  6 months: Type I | 0 | 0 | 0
  6 months: Type II | 17 | 21 | 11
  6 months: Type III | 1 | 0 | 0
  6 months: Type IV | 3 | 1 | 0
  6 months: Type V | 21 | 18 | 7
  6 months: Indeterminate | 0 | 0 | 0
  12 months: number analyzed (Participants) | 13 | 9 | 0
  12 months: Type I | 0 | 0 |
  12 months: Type II | 6 | 3 |
  12 months: Type III | 0 | 0 |
  12 months: Type IV | 2 | 1 |
  12 months: Type V | 5 | 5 |
  12 months: Indeterminate | 0 | 0 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Type I | 0 | 0 |
  24 months: Type II | 1 | 1 |
  24 months: Type III | 0 | 0 |
  24 months: Type IV | 1 | 0 |
  24 months: Type V | 0 | 1 |
  24 months: Indeterminate | 0 | 0 |

17. Secondary Outcome: MRI Tendon Findings: Infraspinatus Sugaya Score
Description: The Sugaya Score was used to determine postoperative cuff integrity of the infraspinatus tendon through magnetic resonance imaging (MRI). Participants were classified as Type I, Type II, Type III, Type IV, Type V, or Indeterminate. Type I indicated sufficient thickness with homogenously low intensity. Type II indicates sufficient thickness with partial high intensity. Type III indicates insufficient thickness without discontinuity. Type IV indicates presence of a minor discontinuity, suggesting a small full-thickness tear. Type V indicates the presence of a major discontinuity, suggesting a medium or large full-thickness tear.
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 40 | 18
Participants
  3 months: number analyzed (Participants) | 31 | 25 | 9
  3 months: Type I | 1 | 0 | 0
  3 months: Type II | 23 | 20 | 5
  3 months: Type III | 0 | 0 | 0
  3 months: Type IV | 0 | 0 | 0
  3 months: Type V | 7 | 5 | 4
  3 months: Indeterminate | 0 | 0 | 0
  6 months: Type I | 1 | 0 | 0
  6 months: Type II | 27 | 31 | 14
  6 months: Type III | 0 | 0 | 0
  6 months: Type IV | 1 | 0 | 0
  6 months: Type V | 13 | 9 | 4
  6 months: Indeterminate | 0 | 0 | 0
  12 months: number analyzed (Participants) | 13 | 9 | 0
  12 months: Type I | 1 | 0 |
  12 months: Type II | 8 | 6 |
  12 months: Type III | 0 | 0 |
  12 months: Type IV | 0 | 0 |
  12 months: Type V | 4 | 3 |
  12 months: Indeterminate | 0 | 0 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Type I | 0 | 0 |
  24 months: Type II | 2 | 1 |
  24 months: Type III | 0 | 0 |
  24 months: Type IV | 0 | 0 |
  24 months: Type V | 0 | 1 |
  24 months: Indeterminate | 0 | 0 |

18. Secondary Outcome: MRI Tendon Findings: Supraspinatus Goutallier Classification
Description: Goutallier grading for the supraspinatus tendon was used to classify the fatty infiltration of the rotator cuff. The Goutallier classification ranged from Grade 0 to Grade 4. Grade 0 indicated a completely normal muscle without any fatty streaks.
  Grade I indicated some fatty streaks. Grade 2 indicated increased fatty infiltration, but more muscle than fat. Grade 3 indicated equal amounts of fat and muscle. Grade 4 indicated more fat than muscle was present. Participants were classified as one of the following:
  * Grade 0
  * Grade I
  * Grade 2
  * Grade 3
  * Grade 4
  * Unable to assess
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: The safety analysis set (SAF) included participants that received the study device with data collected for the time frame and outcome indicated. No (0) Revision subjects completed the 12 or 24 month visit due to the early termination of the study or withdrawal of subject.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 41 | 39 | 18
Participants
  3 months: number analyzed (Participants) | 30 | 25 | 10
  3 months: Grade 0 | 6 | 3 | 1
  3 months: Grade 1 | 22 | 16 | 8
  3 months: Grade 2 | 2 | 4 | 1
  3 months: Grade 3 | 0 | 1 | 0
  3 months: Grade 4 | 0 | 1 | 0
  3 months: Unable to assess | 0 | 0 | 0
  6 months: Grade 0 | 5 | 5 | 1
  6 months: Grade 1 | 30 | 23 | 15
  6 months: Grade 2 | 6 | 7 | 1
  6 months: Grade 3 | 0 | 2 | 0
  6 months: Grade 4 | 0 | 2 | 1
  6 months: Unable to assess | 0 | 0 | 0
  12 months: number analyzed (Participants) | 13 | 9 | 0
  12 months: Grade 0 | 1 | 1 |
  12 months: Grade 1 | 10 | 4 |
  12 months: Grade 2 | 2 | 2 |
  12 months: Grade 3 | 0 | 1 |
  12 months: Grade 4 | 0 | 1 |
  12 months: Unable to assess | 0 | 0 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Grade 0 | 0 | 1 |
  24 months: Grade 1 | 2 | 0 |
  24 months: Grade 2 | 0 | 0 |
  24 months: Grade 3 | 0 | 1 |
  24 months: Grade 4 | 0 | 0 |
  24 months: Unable to assess | 0 | 0 |

19. Secondary Outcome: MRI Tendon Findings: Infraspinatus Goutallier Classification
Description: Goutallier grading for the infraspinatus tendon was used to classify the fatty infiltration of the rotator cuff. The Goutallier classification ranged from Grade 0 to Grade 4. Grade 0 indicated a completely normal muscle without any fatty streaks.
  Grade I indicated some fatty streaks. Grade 2 indicated increased fatty infiltration, but more muscle than fat. Grade 3 indicated equal amounts of fat and muscle. Grade 4 indicated more fat than muscle was present. Participants were classified as one of the following:
  * Grade 0
  * Grade I
  * Grade 2
  * Grade 3
  * Grade 4
  * Unable to assess
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 40 | 40 | 18
Participants
  3 months: number analyzed (Participants) | 29 | 25 | 10
  3 months: Grade 0 | 3 | 6 | 1
  3 months: Grade 1 | 16 | 13 | 3
  3 months: Grade 2 | 8 | 3 | 5
  3 months: Grade 3 | 2 | 2 | 1
  3 months: Grade 4 | 0 | 1 | 0
  3 months: Unable to assess | 0 | 0 | 0
  6 months: Grade 0 | 3 | 9 | 1
  6 months: Grade 1 | 19 | 19 | 10
  6 months: Grade 2 | 13 | 7 | 6
  6 months: Grade 3 | 4 | 3 | 1
  6 months: Grade 4 | 1 | 2 | 0
  6 months: Unable to assess | 0 | 0 | 0
  12 months: number analyzed (Participants) | 13 | 9 | 0
  12 months: Grade 0 | 1 | 1 |
  12 months: Grade 1 | 7 | 6 |
  12 months: Grade 2 | 4 | 1 |
  12 months: Grade 3 | 1 | 0 |
  12 months: Grade 4 | 0 | 1 |
  12 months: Unable to assess | 0 | 0 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Grade 0 | 0 | 1 |
  24 months: Grade 1 | 1 | 0 |
  24 months: Grade 2 | 1 | 0 |
  24 months: Grade 3 | 0 | 0 |
  24 months: Grade 4 | 0 | 1 |
  24 months: Unable to assess | 0 | 0 |

20. Secondary Outcome: Total Tendon Thickness
Description: Post-operative tendon thickness in millimeters (mm) taken from magnetic resonance imaging (MRI).
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: The safety analysis set (SAF) included participants that received the study device with data collected for the time frame and outcome indicated. No (0) Revision subjects completed the 12 or 24 month visit due to the early termination of the study or withdrawal of subject. No (0) ARCR alone subjects tendon thickness at 24 months could be reported as no data was collected because relevant images were missing, not available, or relevant anatomy not visible in field of view.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 20 | 19 | 8
millimeters (mm)
  3 months: number analyzed (Participants) | 17 | 14 | 4
  3 months | 5.6 (1.4) | 5.4 (1.1) | 6.2 (1.5)
  6 months | 5.9 (1.2) | 5.5 (1) | 5.7 (1.1)
  12 months: number analyzed (Participants) | 7 | 3 | 0
  12 months | 4.9 (1) | 5.5 (0.6) |
  24 months: number analyzed (Participants) | 2 | 0 | 0
  24 months | 5 (0.3) |  |

21. Secondary Outcome: Total Tendon Length
Description: Post-operative tendon length in millimeters (mm) taken from magnetic resonance imaging (MRI).
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 29 | 27 | 11
millimeters (mm)
  3 months: number analyzed (Participants) | 23 | 21 | 2
  3 months | 36.4 (9.3) | 32.6 (11.3) | 40.2 (1.3)
  6 months | 34.7 (9.6) | 33.9 (10.4) | 38.2 (4)
  12 months: number analyzed (Participants) | 8 | 6 | 0
  12 months | 33.6 (10.3) | 29.6 (13) |
  24 months: number analyzed (Participants) | 1 | 2 | 0
  24 months | 49.1 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 19.9 (13.6) |

22. Secondary Outcome: Size of Retear: Area (Anteroposterior [AP] / Mediolateral [ML])
Description: Area of retear in millimeters squared (mm^2) at operation day (Day 0), 3 months, and 6 months taken from magnetic resonance imaging (MRI).
Time Frame: Day 0, 3 months and 6 months
Population: The safety analysis set (SAF) included participants that received the study device with data collected for the time frame and outcome indicated.
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 24 | 16 | 7
millimeters squared (mm^2)
  Day 0 | 1041.7 (482.7) | 1004 (448.5) | 877.1 (218.3)
  3 months: number analyzed (Participants) | 12 | 10 | 6
  3 months | 1173.2 (698.5) | 1099.6 (554.1) | 1158.2 (790.8)
  6 months | 1000.6 (699.2) | 1203.0 (624.3) | 1159.6 (1022.3)

23. Secondary Outcome: Size of Retear: Anteroposterior (AP) Length
Description: Anteroposterior (AP) length of retear in millimeters (mm) at operation day (Day 0), 3 months, and 6 months taken from magnetic resonance imaging (MRI).
Time Frame: Day 0, 3 months and 6 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 24 | 16 | 7
millimeters (mm)
  Day 0 | 32.1 (7.2) | 31.8 (7.4) | 30 (8.2)
  3 months: number analyzed (Participants) | 12 | 10 | 6
  3 months | 29.9 (12.5) | 30.7 (9.8) | 28.1 (14.0)
  6 months | 27.4 (12.1) | 29.9 (10.9) | 26.8 (14.3)

24. Secondary Outcome: Size of Retear: Mediolateral (ML) Length
Description: Mediolateral (ML) length of retear in millimeters (mm) at operation day (Day 0), 3 months, and 6 months taken from magnetic resonance imaging (MRI).
Time Frame: Day 0, 3 months and 6 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 24 | 16 | 7
millimeters (mm)
  Day 0 | 31.7 (8.7) | 31.7 (11.4) | 29.4 (1.5)
  3 months: number analyzed (Participants) | 12 | 10 | 6
  3 months | 36.9 (8.9) | 33.6 (11.4) | 37.6 (11.1)
  6 months | 32.1 (12.8) | 37.1 (13.2) | 38.1 (16.4)

25. Secondary Outcome: Shape of Retear: Operative Visit
Description: Shape of tear at operative visit (Day 0) from magnetic resonance imaging (MRI) for those with re-tear at 6 months. Participants were categorized as one of the following tear shapes:
  * Crescent
  * L Shape
  * Reverse L
  * U Shape
  * Massive/Contracted
  * Unable to Determine
Time Frame: Day 0
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 26 | 24 | 13
Participants
  Crescent | 12 | 8 | 7
  L Shape | 2 | 7 | 0
  Reverse L | 1 | 2 | 2
  U Shape | 6 | 4 | 3
  Massive/Contracted | 5 | 3 | 1
  Unable to Determine | 0 | 0 | 0

26. Secondary Outcome: Shape of Retear: 3 Months, 6 Months, 12 Months, and 24 Months
Description: Shape of retear post-operatively at 3 months, 6 months, 12 months and 24 months from magnetic resonance imaging (MRI). Participants were categorized as one of the following retear shapes:
  * Intact (i.e., no re-tear)
  * Crescent
  * Longitudinal
  * Massive
  * Unable to Determine
Time Frame: 3 months, 6 months, 12 months and 24 months
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 40 | 18
Participants
  3 months: number analyzed (Participants) | 31 | 25 | 10
  3 months: Intact (i.e., no re-tear) | 18 | 14 | 3
  3 months: Crescent | 1 | 2 | 0
  3 months: Longitudinal | 4 | 1 | 2
  3 months: Massive | 8 | 8 | 4
  3 months: Unable to Assess | 0 | 0 | 1
  6 months: Intact (i.e., no re-tear) | 16 | 21 | 10
  6 months: Crescent | 3 | 0 | 1
  6 months: Longitudinal | 5 | 4 | 4
  6 months: Massive | 18 | 14 | 3
  6 months: Unable to Assess | 0 | 1 | 0
  12 months: number analyzed (Participants) | 13 | 9 | 0
  12 months: Intact (i.e., no re-tear) | 5 | 3 |
  12 months: Crescent | 0 | 0 |
  12 months: Longitudinal | 3 | 2 |
  12 months: Massive | 4 | 4 |
  12 months: Unable to Assess | 1 | 0 |
  24 months: number analyzed (Participants) | 2 | 2 | 0
  24 months: Intact (i.e., no re-tear) | 1 | 1 |
  24 months: Crescent | 1 | 0 |
  24 months: Longitudinal | 0 | 0 |
  24 months: Massive | 0 | 1 |
  24 months: Unable to Assess | 0 | 0 |

27. Secondary Outcome: Return to Work Questionnaire
Description: Generic questionnaire at 2 weeks, 6 weeks, 3 months, and 6 months with Yes/No responses for the following questions:
  * Returned to work?
  * Have you been able to return to the job you did before your surgery?
  * Did you feel ready to go back to work physically?
  * Since returning to work, any time off due to shoulder pain or weakness?
  * Since last follow-up visit did you take additional time off due to shoulder pain/weakness?
Time Frame: 2 weeks, 6 weeks, 3 months and 6 months
Population: The full analysis set (FAS) followed the Intent-to-Treat principle that included participants enrolled into the study that attended at least one post-surgery assessment with data collected for the time frame and outcome indicated. Each group with 0 participants analyzed for "Since last follow-up visit did you take additional time off..." question at 2 weeks, 6 weeks, 3 months, & 6 months indicated no responses were provided (i.e., data not collected).
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 25 | 25 | 11
Participants
  2 weeks: Returned to work?: Yes | 7 | 5 | 3
  2 weeks: Returned to work?: No | 18 | 20 | 8
  6 weeks: Returned to work?: number analyzed (Participants) | 16 | 19 | 8
  6 weeks: Returned to work?: Yes | 1 | 3 | 3
  6 weeks: Returned to work?: No | 15 | 16 | 5
  3 months: Returned to work?: number analyzed (Participants) | 15 | 13 | 3
  3 months: Returned to work?: Yes | 3 | 2 | 2
  3 months: Returned to work?: No | 12 | 11 | 1
  6 months: Returned to work?: number analyzed (Participants) | 12 | 23 | 6
  6 months: Returned to work?: Yes | 4 | 14 | 3
  6 months: Returned to work?: No | 8 | 9 | 3
  2 weeks: Have you been able to return to the job you did before your surgery?: number analyzed (Participants) | 7 | 5 | 3
  2 weeks: Have you been able to return to the job you did before your surgery?: Yes | 5 | 2 | 1
  2 weeks: Have you been able to return to the job you did before your surgery?: No | 2 | 3 | 2
  6 weeks: Have you been able to return to the job you did before your surgery?: number analyzed (Participants) | 1 | 3 | 3
  6 weeks: Have you been able to return to the job you did before your surgery?: Yes | 1 | 1 | 2
  6 weeks: Have you been able to return to the job you did before your surgery?: No | 0 | 2 | 1
  3 months: Have you been able to return to the job you did before your surgery?: number analyzed (Participants) | 3 | 2 | 2
  3 months: Have you been able to return to the job you did before your surgery?: Yes | 3 | 1 | 1
  3 months: Have you been able to return to the job you did before your surgery?: No | 0 | 1 | 1
  6 months: Have you been able to return to the job you did before your surgery?: number analyzed (Participants) | 4 | 13 | 3
  6 months: Have you been able to return to the job you did before your surgery?: Yes | 4 | 10 | 3
  6 months: Have you been able to return to the job you did before your surgery?: No | 0 | 3 | 0
  2 weeks: Did you feel ready to go back to work physically?: number analyzed (Participants) | 7 | 5 | 3
  2 weeks: Did you feel ready to go back to work physically?: Yes | 5 | 5 | 2
  2 weeks: Did you feel ready to go back to work physically?: No | 2 | 0 | 1
  6 weeks: Did you feel ready to go back to work physically?: number analyzed (Participants) | 1 | 3 | 3
  6 weeks: Did you feel ready to go back to work physically?: Yes | 1 | 3 | 3
  6 weeks: Did you feel ready to go back to work physically?: No | 0 | 0 | 0
  3 months: Did you feel ready to go back to work physically?: number analyzed (Participants) | 3 | 2 | 2
  3 months: Did you feel ready to go back to work physically?: Yes | 3 | 1 | 2
  3 months: Did you feel ready to go back to work physically?: No | 0 | 1 | 0
  6 months: Did you feel ready to go back to work physically?: number analyzed (Participants) | 4 | 14 | 3
  6 months: Did you feel ready to go back to work physically?: Yes | 4 | 12 | 2
  6 months: Did you feel ready to go back to work physically?: No | 0 | 2 | 1
  2 weeks: Since returning to work, any time off due to shoulder pain or weakness?: number analyzed (Participants) | 7 | 5 | 3
  2 weeks: Since returning to work, any time off due to shoulder pain or weakness?: Yes | 0 | 0 | 0
  2 weeks: Since returning to work, any time off due to shoulder pain or weakness?: No | 7 | 5 | 3
  6 weeks: Since returning to work, any time off due to shoulder pain or weakness?: number analyzed (Participants) | 1 | 3 | 3
  6 weeks: Since returning to work, any time off due to shoulder pain or weakness?: Yes | 0 | 0 | 0
  6 weeks: Since returning to work, any time off due to shoulder pain or weakness?: No | 1 | 3 | 3
  3 months: Since returning to work, any time off due to shoulder pain or weakness?: number analyzed (Participants) | 3 | 2 | 2
  3 months: Since returning to work, any time off due to shoulder pain or weakness?: Yes | 0 | 0 | 0
  3 months: Since returning to work, any time off due to shoulder pain or weakness?: No | 3 | 2 | 2
  6 months: Since returning to work, any time off due to shoulder pain or weakness?: number analyzed (Participants) | 4 | 14 | 3
  6 months: Since returning to work, any time off due to shoulder pain or weakness?: Yes | 0 | 1 | 1
  6 months: Since returning to work, any time off due to shoulder pain or weakness?: No | 4 | 13 | 2
  2 weeks: Since last follow-up visit did you take additional time off due to shoulder pain/weakness?: number analyzed (Participants) | 0 | 0 | 0
  6 weeks: Since last follow-up visit did you take additional time off due to shoulder pain/weakness?: number analyzed (Participants) | 0 | 0 | 0
  3 months: Since last follow-up visit did you take additional time off due to shoulder pain/weakness?: number analyzed (Participants) | 0 | 0 | 0
  6 months: Since last follow-up visit did you take additional time off due to shoulder pain/weakness?: number analyzed (Participants) | 0 | 3 | 1
  6 months: Since last follow-up visit did you take additional time off due to shoulder pain/weakness?: Yes |  | 1 | 0
  6 months: Since last follow-up visit did you take additional time off due to shoulder pain/weakness?: No |  | 2 | 1

28. Secondary Outcome: Return to Work Questionnaire: Reason for Not Getting Back to Work
Description: The reason for not getting back to work was a conditional question asked from the Return to Work Questionnaire. Only participants with a 'No' response to the "Returned to work?" question were asked to provide a reason for not getting back to work from one of the following options:
  * Physical capability
  * Safety
  * Motivation
  * Other
Time Frame: 2 weeks, 6 weeks, 3 months, 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 18 | 20 | 8
Participants
  2 weeks: Physical capability | 12 | 13 | 5
  2 weeks: Safety | 1 | 1 | 1
  2 weeks: Motivation | 0 | 0 | 0
  2 weeks: Other | 5 | 6 | 2
  6 weeks: number analyzed (Participants) | 15 | 15 | 5
  6 weeks: Physical capability | 11 | 12 | 4
  6 weeks: Safety | 1 | 0 | 0
  6 weeks: Motivation | 0 | 1 | 0
  6 weeks: Other | 3 | 2 | 1
  3 months: number analyzed (Participants) | 11 | 10 | 1
  3 months: Physical capability | 7 | 8 | 1
  3 months: Safety | 1 | 0 | 0
  3 months: Motivation | 0 | 0 | 0
  3 months: Other | 3 | 2 | 0
  6 months: number analyzed (Participants) | 8 | 8 | 3
  6 months: Physical capability | 3 | 3 | 2
  6 months: Safety | 1 | 1 | 0
  6 months: Motivation | 0 | 0 | 0
  6 months: Other | 4 | 4 | 1

29. Secondary Outcome: Return to Work Questionnaire: Reason Couldn't Return to Activities
Description: The reason for not returning to the same activities was a conditional question asked from the Return to Work Questionnaire. Only participants with a 'No' response to the "Have you been able to return to the job you did before your surgery?" question were asked to provide a reason for not getting back to work from one of the following options:
  * Physical capability
  * Safety
  * Motivation
  * Other
Time Frame: 2 weeks, 6 weeks, 3 months, 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 2 | 3 | 2
Participants
  2 weeks: Physical capability | 2 | 3 | 2
  2 weeks: Safety | 0 | 0 | 0
  2 weeks: Motivation | 0 | 0 | 0
  2 weeks: Other | 0 | 0 | 0
  6 weeks: number analyzed (Participants) | 0 | 2 | 1
  6 weeks: Physical capability |  | 1 | 1
  6 weeks: Safety |  | 1 | 0
  6 weeks: Motivation |  | 0 | 0
  6 weeks: Other |  | 0 | 0
  3 months: number analyzed (Participants) | 0 | 1 | 1
  3 months: Physical capability |  | 1 | 1
  3 months: Safety |  | 0 | 0
  3 months: Motivation |  | 0 | 0
  3 months: Other |  | 0 | 0
  6 months: number analyzed (Participants) | 0 | 3 | 0
  6 months: Physical capability |  | 2 |
  6 months: Safety |  | 0 |
  6 months: Motivation |  | 0 |
  6 months: Other |  | 1 |

30. Secondary Outcome: Return to Work Questionnaire: Time Off
Description: Number of days taken off after returning to work because of shoulder pain or weakness was a conditional question asked from the Return to Work Questionnaire. Only participants with a 'Yes' response to the "Since returning to work, any time off due to shoulder pain or weakness?" question were asked to provide how long they have taken off in days.
Time Frame: 2 weeks, 6 weeks, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 0 | 1 | 1
days
  2 weeks: number analyzed (Participants) | 0 | 0 | 0
  6 weeks: number analyzed (Participants) | 0 | 0 | 0
  3 months: number analyzed (Participants) | 0 | 0 | 0
  6 months |  | 8 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 2 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis

31. Secondary Outcome: Return to Work Questionnaire: Duration Away From Work (Days)
Description: Number of days taken away from work following surgery was a conditional question asked from the Return to Work Questionnaire. Only participants with a 'Yes' response to the "Returned to work?" question were asked to provide the number of days taken away from work
Time Frame: 2 weeks, 6 weeks, 3 months, 6 months
Population: The full analysis set (FAS) followed the Intent-to-Treat principle that included participants enrolled into the study that attended at least one post-surgery assessment with data collected for the time frame and outcome indicated. Data not collected for 2 subjects who responded yes at 6 months in ARCR alone group.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 7 | 12 | 3
days
  2 weeks: number analyzed (Participants) | 7 | 5 | 3
  2 weeks | 6.7 (3) | 7.2 (4.4) | 6.7 (5.1)
  6 weeks: number analyzed (Participants) | 1 | 3 | 3
  6 weeks | 19 (NA) — Standard Deviation could not be calculated because only 1 participant had data collected for analysis | 23 (4.6) | 30.3 (15.9)
  3 months: number analyzed (Participants) | 3 | 2 | 2
  3 months | 68.3 (20.8) | 64.5 (16.3) | 52 (11.3)
  6 months: number analyzed (Participants) | 4 | 12 | 3
  6 months | 74.5 (69.9) | 80.3 (63.8) | 75 (18.7)

32. Secondary Outcome: Duration of Opioid Use
Description: Duration of opioid use in days up to 14 days post-surgery was based on self-reported opioid use diary completed by the patient on a daily basis for 2 weeks after surgery.
Time Frame: Following surgery, up to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 42 | 21
days | 7.9 (4.9) | 7.1 (4.5) | 6.3 (4.9)

33. Secondary Outcome: Opioid Use for More Than 5 Days Post-Surgery
Description: Number of participants taking opioids for more than 5 days post-surgery (Yes/No) was based on self-reported opioid use diary completed by the patient on a daily basis for 2 weeks after surgery.
Time Frame: Following surgery, up to 14 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 42 | 42 | 21
Participants
  No | 17 | 18 | 10
  Yes | 25 | 24 | 11

34. Secondary Outcome: Total Operative Time
Description: Total operative time in minutes.
Time Frame: Intraoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 46 | 48 | 24
minutes | 176.2 (60.9) | 138.8 (42.7) | 172.8 (47.7)

35. Secondary Outcome: Sling Type
Description: The type of sling used up to 3 months post-surgery for each participant was categorized as one of the following:
  * Standard Sling
  * Shoulder Immobilizer
  * Sling and Swathe
  * Abduction Sling
  * External Rotation Sling
  * Other
  * Missing
Time Frame: up to 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 46 | 48 | 24
Participants
  Standard Sling | 13 | 17 | 5
  Shoulder Immobilizer | 20 | 16 | 6
  Sling and Swathe | 0 | 0 | 0
  Abduction Sling | 8 | 4 | 4
  External Rotation Sling | 0 | 3 | 0
  Other | 4 | 4 | 7
  Missing | 1 | 4 | 2

36. Secondary Outcome: Mobilization Time in Sling
Description: Mobilization time was the duration, measured in weeks, that participants spent in a sling.
Time Frame: up to 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
Number analyzed (Participants) | 45 | 45 | 22
weeks | 5.5 (1.1) | 5.4 (1.3) | 5.6 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during surgery to early termination, up to 24 months.
Arm/Group | ARCR Augmented With REGENETEN™ Bioinductive Implant | ARCR Alone | Revision Group
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/47 | 6/48 | 4/24
Other Adverse Events (participants affected / at risk) | 16/47 | 11/48 | 4/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARCR Augmented With REGENETEN™ Bioinductive Implant (N=47) | ARCR Alone (N=48) | Revision Group (N=24)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
Stroke/CVA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
Low Blood Pressure/Hypotension (General disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to device
Syncope/Fainting (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to device
Loss of Range of Motion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
Muscle/Tendon Damage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to device
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Unrelated to device
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Unrelated to device
Muscle/Tendon Damage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Serious adverse device effect. Unrelated to device, definite relationship to study procedure
Muscle/Tendon Damage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Serious adverse device effect. Unrelated to device, possible relationship to study procedure
Loss of Range of Motion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Serious adverse device effect. Unrelated to device, possible relationship to study procedure
Unspecified Musculoskeletal Problem (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Serious adverse device effect. Unrelated to device, definite relationship to study procedure
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — Serious adverse device effect. Possible relationship to device, possible relationship to study procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARCR Augmented With REGENETEN™ Bioinductive Implant (N=47) | ARCR Alone (N=48) | Revision Group (N=24)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (2)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Nervous Injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Unspecified Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling/Edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Post Operative Wound Infection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sleep Dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Low Oxygen Saturation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Insufficient Information (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Damage to Ligament(s) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin Inflammation/Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 1 (1) — Adverse device effect. Possible relationship to device and study procedures.
Pain (General disorders) | 1 (2) | 1 (1) | 1 (1) — Adverse device effect. Unrelated to device, possible relationship to study procedures.
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Adverse device effect. Unrelated to device, possible relationship to study procedures.
Hemorrhage/Bleeding (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Adverse device effect. Unrelated to device, definite relationship to study procedures.
Loss of Range of Motion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Adverse device effect. Unrelated to device, definite relationship to study procedures.
Swelling/Edema (General disorders) | 2 (2) | 1 (1) | 0 (0) — Adverse device effect. Unrelated to device, possible relationship to study procedures.
Unspecified Musculoskeletal Problem (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Adverse device effect. Unrelated to device, definite relationship to study procedures.
Foreign Body in Patient (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Adverse device effect. Definite relationship to device and study procedures.
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Adverse device effect. Unrelated to device, possible relationship to study procedures.
Unspecified Musculoskeletal Problem (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Adverse device effect. Unrelated to device, possible relationship to study procedures.
Swelling/Edema (General disorders) | 1 (1) | 0 (0) | 0 (0) — Adverse device effect. Unrelated to device, definite relationship to study procedures.
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Adverse device effect. Unrelated to the device, possible relationship to study procedures. Sponsor disagreed with this classification (believed it to be an adverse event) however the most stringent classification has been reported.

LIMITATIONS AND CAVEATS:
The study was terminated early (Sponsor decision not related to safety) following completion the 6-month follow-up visit due to the numerous risk factors for re-tear, such as tear size and tendon medialization. The number and variability of risk factors present made it impractical to achieve a sample size necessary to statistically account for all risk factors and evaluate the influence of augmentation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon completion of the Trial the PI may prepare the data derived from the Trial for publication, and will submit to Sponsor for review and comment prior to publication. To ensure that Sponsor will be able to make comment and suggestions where pertinent, the material for public dissemination will be submitted for review at least 40 to 90 days* prior to submission for publication, public dissemination or review by a publication committee.

*Country dependent, no timeframe is mandated for France.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT04450342/Prot_SAP_000.pdf